CLINICAL TRIAL: NCT00416611
Title: IMPlementation of gUideLines for the Management of Arterial hypertenSION. The IMPULSION Study
Acronym: IMPULSION
Status: Completed | Type: Observational
Sponsor: Hellenic Atherosclerosis Society (Other)
Responsible Party: Hellenic Atherosclerosios Society, V. Athyros, MD member of Advisdory Board of Hellenic Atherosclerosios Society
Other Study IDs: HAS-02-231206
Record Dates: First submitted 2006-12-23; First posted 2006-12-28 (Estimated); Last update posted 2009-01-29 (Estimated); Status verified 2009-01

CONDITIONS: High Blood Pressure
Keywords: High blood pressure; Awareness; Treatment; Effective Control; Coronary heart disease risk reduction; Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Behavioral: Implementation of guidelines

SUMMARY:
The objective of this protocol is to improve awareness, treatment, and control of arterial hypertension, within primary prevention of target organ damage, by implementing guidelines, after training of the participating physicians.

DETAILED DESCRIPTION:
Physicians from 20 hospitals and 40 health centres (primary health care settings) were trained to implement guidelines in treating arterial hypertension.

There will be a baseline recording of patients with arterial hypertension and then physicians will have to complete a one page form (by ticking pre-specified boxes) about the baseline status of the patients and will have to report the measures they took to improve awareness, treatment, and effective control of arterial hypertension. After a six month effort, physicians will have to complete the same form at study completion. Previous training of physicians and the fact that they will have to report their success in treating hypertension will hopefully contribute to an increase in number of hypertensive patients at blood pressure target, and will minimise the target organ damage. The estimated reduction in coronary heart disease risk will be evaluated by a comparison of this risk (as evaluated by a risk engine, i.e. PROCAM) at study completion with that of baseline.

ELIGIBILITY:
Inclusion Criteria:

* Arterial hypertension as defined by the JNC 7 report

Exclusion Criteria:

* Pregnancy
* Lactation
* Malignancies with small life expectancy
* Unwillingness to participate

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2006-11; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Efficacy in arterial hypertension control | 6 months
Efficacy in reducing estimated risk of coronary heart disease | 6 months

SECONDARY OUTCOMES:
Cost effectiveness of arterial hypertension control | 6 months
Differences between primary and secondary health care settings as well as teaching hospitals | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Athyros G Athyros, MD, Study Director — Clinical Trials Chair of Hellenic Atherosclerosis Society
Locations (1):
- Hellenic Atherosclerosis Society, Thessaloniki, Thessaloniki, Greece

REFERENCES:
- [Result] Karagiannis A, Athyros VG, Papageorgiou A, Tziomalos K, Elisaf M. Should atenolol still be recommended as first-line therapy for primary hypertension? Hellenic J Cardiol. 2006 Sep-Oct;47(5):298-307. No abstract available. PMID 17134065
- [Derived] Karagiannis A, Hatzitolios AI, Athyros VG, Deligianni K, Charalambous C, Papathanakis C, Theodosiou G, Drakidis T, Chatzikaloudi V, Kamilali C, Matsiras S, Matziris A, Savopoulos C, Baltatzi M, Rudolf J, Tziomalos K, Mikhailidis DP. Implementation of guidelines for the management of arterial hypertension. The impulsion study. Open Cardiovasc Med J. 2009 May 5;3:26-34. doi: 10.2174/1874192400903010026. PMID 19557149